CLINICAL TRIAL: NCT02498587
Title: Short Period Incidence Study of Severe Acute Respiratory Illness
Acronym: SPRINT-SARI
Status: Recruiting | Type: Observational
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: International Severe Acute Respiratory and Emerging Infection Consortium (Other); The International Forum of Acute Care Trialists (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANZIC-RC/SW0002
Record Dates: First submitted 2015-03-26; First posted 2015-07-15 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Severe Acute Respiratory Infection
Keywords: Severe Acute Respiratory Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-centre, prospective, short period incidence observational study of patients in participating hospitals and intensive care units (ICUs) with SARI. The study period will occur, in both Northern and Southern hemispheric winters. The study period will comprise a 5 to 7-day cohort study in which patients meeting a SARI case-definition, who are newly admitted to the hospitals / ICUs at participating sites, will be included in the study. The study will be conducted in 20 to 40-hospital/ ICU-based research networks globally. All clinical information and sample data will only be recorded if taken as part of the routine clinical practice at each site and only fully anonymised and de-identified data will be submitted centrally.

The primary aim of this study is to establishing a research response capability for a future epidemic / pandemic through a global SARI observational study. The secondary aim of this study is to investigate the descriptive epidemiology and microbiology profiles of patients with SARI. The tertiary aim of this study is to assess the Ethics, Administrative, Regulatory and Logistic (EARL) barriers to conducting pandemic research on a global level.

DETAILED DESCRIPTION:
Severe acute respiratory infection (SARI) continues to be of major relevance to public health worldwide. In the last 10 years there have been multiple SARI outbreaks around the world. The 2009 H1N1 pandemic was estimated to result in more than 200,000 respiratory deaths globally. The World Health Organization (WHO) defines SARI as an acute respiratory infection of recent onset (within 10 days) requiring hospitalisation, manifested by fever (≥38oC) or a history of fever and cough. There is international consensus that it is important to undertake observational studies of patients with SARI as an essential component of pandemic and epidemic research preparedness.

ELIGIBILITY:
Inclusion Criteria:

* A history of feverishness or measured fever of ≥ 38 deg C;
* Cough;
* Dyspnoea (shortness of breath) OR Tachypnoea.

Exclusion Criteria:

• No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients newly admitted to participating hospitals, of any age, presenting with SARI during the study period. Patients will be eligible for the study if the patient meets the case definition for SARI.
  A suspected or proven acute respiratory infection requiring new inpatient admission with onset within the past 14 days. With one or more of the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participating sites | one week
  The number of sites able to participate and submit data for central analysis
Data Completeness | 90 days
  The completeness of submitted data
Barriers to data submission | 90 days
  Survey post SPRINT-SARI study period on barriers to data completion

SECONDARY OUTCOMES:
Incidence of SARI | one week
  Number of participants during the study period at all sites
Length of Hospital Stay | 90 days
  Length of stay of SARI patients by co-morbidities and risk factors
Symptoms at admission | 90 days
  Impact of different SARI case definitions on cohort
Incidence of Intensive Care Unit Admission | 90 days
  Rate of ICU admission in SARI cohorts and international variation
Length of Intensive Care Unit Admission | 90 days
  Length of stay for participants admitted to an ICU during SARI hospital admission
SARI Microbiology | 90 days
  Microbiological SARI diagnosis of participants (if known) during hospital admission

OTHER OUTCOMES:
Global Ethical Approval requirements | 90 days
  Survey post SPRINT-SARI study period of ethical approval requirements in participating countries
Time requirements for obtaining Ethical approval | 90 days
  Survey post SPRINT-SARI study period of time required to obtain ethical approval for SPRINT-SARI at participating sites

CONTACTS AND LOCATIONS:
Locations (1):
- Australian and New Zealand Intensive Care Research Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes